CLINICAL TRIAL: NCT04940182
Title: A Multicenter, Adaptive, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of XC221, Tablets, 100 mg in Patients With Mild COVID-19
Brief Title: A Study to Assess the Efficacy and Safety of XC221 in Patients With Mild COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RSV Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XC221-03-03-2020
Record Dates: First submitted 2021-06-23; First posted 2021-06-25 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Sars-CoV-2 Infection
Keywords: COVID-19; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — XC221

STUDY DESIGN:
Intervention Model Description: Two groups (Group A and Group B) in a 1:1 ratio: Group A - investigational product; Group В - Placebo.
Who Masked: Participant, Investigator
Masking Description: Tablets identical in terms of composition, appearance and labeling to XC221 tablets, but without active substance will be used as Placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XC221 (Experimental): XC221 100 mg orally. 1 tablet of XC221 100 mg 2 times a day during 14 full days of treatment period
  Interventions: Drug: XC221
- Placebo (Placebo Comparator): Placebo orally. 1 tablet of Placebo 2 times a day during 14 full days of treatment period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XC221 — Participants will receive XC221 100 mg 2 times a day during 14 full days
  Arms: XC221
Drug: Placebo — Participants will receive Placebo 2 times a day during 14 full days
  Arms: Placebo

SUMMARY:
The innovative drug XC221 100 mg tablet is designed for the treatment of COVID-19 (SARS-CoV-2 infection). A multicenter, adaptive, randomized, double-blind, placebo-controlled Phase III clinical study is aimed to assess the efficacy and safety of XC221 100 mg tablet, in mild COVID-19 patients during a 14-days treatment.

The primary objective of the study is to demonstrate the efficacy of XC221 100 mg tablet (200 mg daily dose) in achieving clinical improvement of mild COVID-19 symptoms.

The secondary objective of the study is to evaluate the safety of XC221 100 mg tablet (200 mg daily dose) in mild COVID-19 patients.

DETAILED DESCRIPTION:
8 Russian centers will participate in this study. The trail will consist of three periods: screening (duration not more than 1 day, it may coincide with the randomization visit and beginning of drug administration), treatment period (14 full days) and follow-up period (15 ± 1 days after completion of treatment with XC221 / Placebo). The duration of participation in the study for each patient will be no more than 32 days.

274 eligible patients with confirmed COVID-19 will be randomized into two groups (Group A and Group B) in a 1:1 ratio: Group A - XC221 200 mg daily (137 patients); Group В - Placebo (137 patients).

During the treatment period (14 full days), 1 tablet of XC221 / Placebo will be administered 2 times a day in addition to the standard of care (SoC) for COVID-19 according to The Temporary guidelines for the prevention, diagnosis and treatment of SARS-CoV-2 infection of the Ministry of Health of the Russian Federation (the MoH Temporary Guidelines). The follow-up period will last for 15 ± 1 days.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form.
2. Patients of both sexes aged 18 to 75 years inclusive.
3. Diagnosed COVID-19 based on positive laboratory tests confirming the SARS-CoV-2 presence, performed no earlier than 3 days before screening. It is allowed to determine the SARS-CoV-2 by the PCR or by another method according to the MoH Temporary Guidelines.
4. Patients having a total score ≥ 5 according to the COVID-19 Major Symptom Rating Scale.
5. Patients with mild COVID-19, as defined in The MoH Temporary Guidelines. Presence of at least two criteria: SpO2 ≥ 95% (required criterion), 37.5°С ≤ t ˂ 38°С, or respiratory rate (RR) ≤ 22 / min. Absence of moderate/severe progression criteria.
6. Disease duration is no more than 3 full days since the onset of one or more of symptoms below before the first dose of the drug administration:

   * body temperature increase;
   * dry cough or cough with little phlegm;
   * dyspnoea;
   * myalgia;
   * fatigue;
   * feeling of congestion in the chest;
   * reduced sense of smell and / or taste.
7. For women only: negative pregnancy test result. Pregnancy testing is not required for women of not childbearing potential (WONCBP): women who are in menopause (defined as an absence of menstruation for at least 2 years or more), or women who undergone surgical sterilization (hysterectomy, bilateral oophorectomy, tubal ligation), or women with a clinical diagnosis of "infertility". The presence of surgical sterilization and infertility should be confirmed by patient's claim or by relevant document confirming this condition.
8. Consent to use reliable method of contraception throughout the study period.
9. Patients who are able to understand and comply with treatment and procedures during the study.

Exclusion Criteria:

1. Known or suspected hypersensitivity to the active substance or to excipients of the drug XC221 or placebo
2. Known or suspected hypersensitivity to standard therapy drugs specified in The MoH Temporary Guidelines.
3. Body temperature ˂37.5°С.
4. Lactase deficiency, lactose intolerance, glucose-galactose malabsorption.
5. Presence or suspicion of oncological diseases by the day of criteria assessment or in medical history (within the last 2 years).
6. Presence of autoimmune diseases by the day of criteria assessment or in medical history.
7. Pregnancy.
8. Lactation period.
9. Presence of serious lung diseases, including, but not limited to the following diseases: moderate and severe bronchial asthma, severe and extremely severe COPD, interstitial lung disease, pulmonary hypertension, pulmonary fibrosis, surgical interventions on the lungs, tuberculosis (including suspicion of tuberculosis based on the results of CT examination at screening).
10. Patients with type 1 diabetes mellitus and / or decompensated type 2 diabetes mellitus.
11. Heart failure, NYHA functional class III - IV.
12. Chronic liver failure stage II (decompensated) and higher.
13. The need of replacement renal therapy at enrollment.
14. Organ transplantation in medical history.
15. Medical history of epilepsy or the need for anticonvulsant therapy.
16. Major depressive disorder, anxiety, other mental disorders requiring medical correction.
17. Acute cerebrovascular accident, stroke or transient ischemic attack within 90 days before screening.
18. Use of any antiviral and / or immunomodulatory drugs after the manifestation of COVID-19.
19. Any immunosuppressive therapy (including tocilizumab / sarilumab) within 90 days prior to randomization, or the need of immunosuppressive therapy at the time of randomization.
20. Use of anti-COVID-19 plasma within 14 days prior to the screening visit.
21. Use of systemic glucocorticosteroids within 90 days prior to randomization, or the need of systemic glucocorticosteroids at the time of randomization.
22. Use of vaccines against viral infections within 90 days prior to randomization.
23. Patients receiving other experimental drugs, drugs not approved in the Russian Federation, or participating in other clinical trials within 30 days before screening.
24. Patients abusing alcohol or psychotropic drugs and other drugs by the day of criteria assessment or during the last year.
25. Patients with other serious, unstable, or clinically significant medical or psychological conditions that, in the opinion of the investigator, may preclude the patient's participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2021-06-26 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Total incidence frequency of progression to moderate COVID-19 illness or worse throughout the study (by Day 31) | Day 1 - Day 31
  Moderate illness parameters:
  * Body temperature > 37.5°C;
  * RR > 22 / min;
  * Dyspnea during exercise;
  * Changes in CT (X-Ray) typical of viral disease (the volume of affected area is minimal or medium, CT 1-2);
  * SpO2 ˂ 95%;
  * Serum CRP > 10 mg/l For the symptoms (body temperature, RR, dyspnea during exercise, SpO2, progression to moderate COVID-19 or worse), the presence of moderate progression criteria as shown by the second of two consecutive measurements.
The median time to a stable decrease in the total score on the COVID-19 Major Symptom Rating Scale to ≤ 1. A stable total score decrease is the presence of 1 point or less as shown by the second of two consecutive measurements | Day 1 - Day 31
  The COVID-19 Major Symptom Rating Scale will be used to assess the individuals' subjective ratings the severity of 9 symptoms of COVID-19. Ranges for each symptom: 0 points (no symptoms) - 3 points (the most severe). Total score (ranges from 0 to 27 points) is a sum of points for each symptom.

SECONDARY OUTCOMES:
Patient rate with improvement for one or more grades of the WHO Scale by Day 2-31 | Day 1 - Day 31
  The scale of the patient's clinical condition, proposed by the WHO, will be used to assess the severity of patient general condition. Ranges for patient's clinical condition: 0 points (no infection) - 8 points (death).
Patient rate with worsening for one or more grades of the WHO Scale by Day 2-31 | Day 1 - Day 31
  The scale of the patient's clinical condition, proposed by the WHO, will be used to assess the severity of patient general condition. Ranges for patient's clinical condition: 0 points (no infection) - 8 points (death).
Mean WHO Scale grade changes from baseline by Day 2-31 | Day 1 - Day 31
  The scale of the patient's clinical condition, proposed by the WHO, will be used to assess the severity of patient general condition. Ranges for patient's clinical condition: 0 points (no infection) - 8 points (death).
Patient rate with SpO2 ≤ 93% by Day 2-31 | Day 1 - Day 31
Patient rate with SpO2 ˂ 95% by Day 2-31 | Day 1 - Day 31
Mean change from baseline in SpO2 by Day 2-31 | Day 1 - Day 31
Patient rate with RR > 22/min by Days 3, 6, 9, 12 and 15 | Day 1 - Day 15
Patient rate with RR > 30/min by Days 3, 6, 9, 12 and 15 | Day 1 - Day 15
Patient rate with RR ≤ 20/min by Days 3, 6, 9, 12 and 15 | Day 1 - Day 15
Mean change from baseline in RR by Days 3, 6, 9, 12 and 15 | Day 1 - Day 15
Patient rate with a body temperature ≤ 37.0°С by Day 2-31 | Day 1 - Day 31
Patient rate with a body temperature ≤ 37.5°С by Day 2-31 | Day 1 - Day 31
Patient rate with a body temperature ≥ 38.5°С by Day 2-31 | Day 1 - Day 31
Mean change from baseline in body temperature by Day 2-31 | Day 1 - Day 31
Patient rate with a score ≤ 1 according to the Daytime and Nighttime Cough Scale by Day 2-31 | Day 1 - Day 31
Mean score change from baseline in the Daytime and Nighttime Cough Scale by Day 2-31 | Day 1 - Day 31
  The Daytime and Nighttime Cough Scale will be used to assess the dynamics of cough during the study. Ranges for assess: 0 points (no cough) - 5 points (cough that prevents sleep).
Average time to reach ≤ 1 score according to the Daytime and Nighttime Cough. | Day 1 - Day 31
  The Daytime and Nighttime Cough Scale will be used to assess the dynamics of cough during the study. Ranges for assess: 0 points (no cough) - 5 points (cough that prevents sleep).
Patient rate with decrease for one or more grades for each symptom according to the COVID-19 Major Symptom Rating Scale by Day 2-31 | Day 1 - Day 31
  The COVID-19 Major Symptom Rating Scale will be used to assess the individuals' subjective ratings the severity of 9 symptoms of COVID-19. Ranges for each symptom: 0 points (no symptoms) - 3 points (the most severe). Total score (ranges from 0 to 27 points) is a sum of points for each symptom.
Patient rate with clinical improvement (1 point or less) for each symptom according to the COVID-19 Major Symptom Rating Scale | Day 1 - Day 31
  The COVID-19 Major Symptom Rating Scale will be used to assess the individuals' subjective ratings the severity of 9 symptoms of COVID-19. Ranges for each symptom: 0 points (no symptoms) - 3 points (the most severe). Total score (ranges from 0 to 27 points) is a sum of points for each symptom.
Time till clinical improvement (1 point or less) for each symptom according to the COVID-19 Major Symptom Rating Scale | Day 1 - Day 31
  The COVID-19 Major Symptom Rating Scale will be used to assess the individuals' subjective ratings the severity of 9 symptoms of COVID-19. Ranges for each symptom: 0 points (no symptoms) - 3 points (the most severe). Total score (ranges from 0 to 27 points) is a sum of points for each symptom.
Patient rate with a grade ≤ 1 for each symptom according to the COVID-19 Major Symptom Rating Scale by Day 2-31 | Day 1 - Day 31
  The COVID-19 Major Symptom Rating Scale will be used to assess the individuals' subjective ratings the severity of 9 symptoms of COVID-19. Ranges for each symptom: 0 points (no symptoms) - 3 points (the most severe). Total score (ranges from 0 to 27 points) is a sum of points for each symptom.
Mean score change from baseline for each symptom according to the COVID-19 Major Symptom Rating Scale by Day 2-31 | Day 1 - Day 31
  The COVID-19 Major Symptom Rating Scale will be used to assess the individuals' subjective ratings the severity of 9 symptoms of COVID-19. Ranges for each symptom: 0 points (no symptoms) - 3 points (the most severe). Total score (ranges from 0 to 27 points) is a sum of points for each symptom.
Average time to reach ≤ 1 score for each symptom according to the COVID-19 Major Symptom Rating Scale | Day 1 - Day 31
  The COVID-19 Major Symptom Rating Scale will be used to assess the individuals' subjective ratings the severity of 9 symptoms of COVID-19. Ranges for each symptom: 0 points (no symptoms) - 3 points (the most severe). Total score (ranges from 0 to 27 points) is a sum of points for each symptom.
Patient rate with a grade ≤ 1 according to the Dyspnea Visual Analogue Scale by Day 2-31 | Day 1 - Day 31
  The Dyspnea Visual Analogue Scale will be used to assess the severity of dyspnea. The scale has five numerical values, rated from 0 (no shortness of breath) to 4 (very severe shortness of breath).
Mean score change from baseline according to the Dyspnea Visual Analogue Scale by Day 2-31 | Day 1 - Day 31
  The Dyspnea Visual Analogue Scale will be used to assess the severity of dyspnea. The scale has five numerical values, rated from 0 (no shortness of breath) to 4 (very severe shortness of breath).
Average time to reach ≤ 1 score according to the Dyspnea Visual Analogue Scale | Day 1 - Day 31
  The Dyspnea Visual Analogue Scale will be used to assess the severity of dyspnea. The scale has five numerical values, rated from 0 (no shortness of breath) to 4 (very severe shortness of breath).
Patient rate with a negative SARS-CoV-2 test result by Day 3, 9, 15, also by Day 7 and Day 15 after the end of drug administration (in the case of a positive previous test result) | Day 1 - Day 31
Time till elimination SARS-CoV-2 | Day 1 - Day 31
Mean CRP concentration change from baseline by Day 15 | Day 1 - Day 15

CONTACTS AND LOCATIONS:
Locations (11):
- Russia (11):
  - Municipal Budgetary Institution of Healthcare "Central City Hospital of Novoshakhtinsk", Novoshakhtinsk, Rostov Oblast
  - Regional Budgetary Institution of Healthcare "Ivanovskaya Clinical Hospital named after Kuvaevykh", Ivanovo
  - State Budgetary Institution of Healthcare of Moscow "City Polyclinic No. 2 of the Moscow Department of Healthcare", Moscow
  - Federal Budgetary Institution of Science "Moscow Research Institute of Epidemiology and Microbiology named after G.N. Gabrichevsky" of the Federal Service for the Oversight of Consumer Protection and Welfare, Moscow
  - Limited Liability Company "Medical Center "Capital-Policy", Saint Petersburg
  - Limited Liability Company "Research Center Eco-Safety", Saint Petersburg
  - LLC "Sphere-Med", Saint Petersburg
  - Saint Petersburg State Budgetary Institution of Healthcare "City Pokrovskaya Hospital" (4th Cardiology Department), Saint Petersburg
  - Saint Petersburg State Budgetary Institution of Healthcare "City Polyclinic No. 4", Saint Petersburg
  - Regional State Budgetary Institution of Healthcare "Medical-Sanitary Unit No. 2", Tomsk
  - LLC "Family Clinic", Yekaterinburg

IPD SHARING:
Plan to Share IPD: No